CLINICAL TRIAL: NCT04740788
Title: Multicentric Retrospective/Prospective Study on Visual Performance of a Monofocal Intraocular Lens (IOL)
Brief Title: Study on Visual Performance of a Monofocal Intraocular Lens
Status: Completed | Type: Observational
Sponsor: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Other Study IDs: GPAS-SUR-020-02
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Cataract Senile

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Monofocal IOL: Patients already implanted with a monofocal IOL
  Interventions: Device: Monofocal IOL

INTERVENTIONS:
Device: Monofocal IOL — Patients are already implanted with a monofocal lens

SUMMARY:
Retrospective/Prospective Study on Visual Performance of a Monofocal Intraocular Lens (IOL). The objective is to compare best corrected distance visual acuity (CDVA) between 1-3-month and 12- month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older;
* Patients with monolateral or bilateral (only one eye will be the study eye) monofocal IOL implantation after uncomplicated surgery in the period between May 2019 and November 2019, if the follow-up visit can be performed 10-18 months after surgery;
* No visual acuity limiting pathologies;
* Availability of 1-3-month postoperative data
* Availability, willingness and sufficient cognitive awareness to comply with examination procedures in case of a prospective 12-month visit;
* Written informed consent for participation in the study and data protection.

Exclusion Criteria:

* Difficulty for cooperation (distance from their home, general health conditions)
* Subjects with diagnosed degenerative visual disorders (e.g. macular degeneration or other retinal or optic disorders) that would confound visual acuity measurements;
* Subjects with surgical complications or secondary interventions (except for Nd:YAG capsulotomy) related to the cataract surgery of the monofocal IOL eye(s) or any other interventions in the post-operative eye including but not limited to glaucoma surgery, retinal surgery;
* Visual field loss which has impact on visual acuity;
* Use of systemic or ocular medication that might affect vision;
* Patients with amblyopia, strabismus, forme fruste keratoconus or keratoconus;
* Capsular or zonular abnormalities that have affected postoperative centration or tilt of the lens (e.g. pseudoexfoliation syndrome);
* Concurrent participation in another device investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cataract patients already implanted with a monofocal IOL
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
Best corrected distance visual acuity (CDVA) | 12 months
  Comparison between 1-3-month and 12- month follow-up results.

CONTACTS AND LOCATIONS:
Locations (1):
- Borkenstein & Borkenstein, Graz, Austria